CLINICAL TRIAL: NCT03256305
Title: A Clinical Control Study of rTMS Personalized Precision Treatment of Post-stroke Depression Based on Mechanism of Emotional Circuit Imbalance
Brief Title: A Study of rTMS Personalized Precision Treatment of Post-stroke Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-KFYXK-001
Record Dates: First submitted 2017-07-18; First posted 2017-08-22 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2017-08

CONDITIONS: Post-stroke Depression
Keywords: Repetitive transcranial magnetic stimulation

STUDY DESIGN:
Intervention Model Description: Care Provider, Investigator, Outcomes Assessor
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- "personalized" rTMS+drug treatment (Experimental): Received "personalized" rTMS treatment 15 times for 15 days;Take paroxetine for 2 weeks
  Interventions: Device: "personalized" rTMS+drug treatment
- Traditional rTMS +drug treatment (Active Comparator): Received traditional rTMS treatment 15 times for 15 days;Take paroxetine for 2 weeks
  Interventions: Device: Traditional rTMS +drug treatment

INTERVENTIONS:
Device: "personalized" rTMS+drug treatment — High frequency（10HZ）stimulation of brain regions corresponding to lesion, low-frequency （1HZ）stimulation of the contralateral brain, intensity=90%MT（motor thresholds). Each sequence is 20 times, duration is 10 seconds, each sequence spaced 60s, 20 sequences per day, 1 times a day ,total times is 15. Taking paroxetine 2 weeks, Take 20 mg a day.
  Other Names: P rTMS
  Arms: "personalized" rTMS+drug treatment
Device: Traditional rTMS +drug treatment — Traditional rTMS treatment protocol parameters: localization of left DLPFC: frequency=10 Hz; localization of right DLPFC: frequency=1 Hz, intensity=90%MT, Each sequence is 20 times, duration is 10 seconds, each sequence spaced 60s, 20 sequences per day,1 times a day,total times is 15. Taking paroxetine 2 weeks, Take 20 mg a day.
  Other Names: T rTMS
  Arms: Traditional rTMS +drug treatment

SUMMARY:
This is a multicenter, randomized trial aims to reveal the efficacy and safety of Repetitive transcranial magnetic stimulation (rTMS) individualized therapy based on the 'emotional loop destabilization' mechanism of PSD .One hundred and twenty participants will be recruited from three centers and randomized with a 1:1 ratio to receive "Personalized" rTMS treatment or traditional rTMS treatment in addition to routine antidepressant treatments.The data of neuropsychological tests and MRI will be collected at 0, 2，4 and 8 weeks after the commencement of the treatment.

DETAILED DESCRIPTION:
This is a multicenter, randomized trial aims to reveal the efficacy and safety of rTMS individualized therapy based on the 'emotional loop destabilization' mechanism of PSD .One hundred and twenty participants will be recruited from three centers and randomized with a 1:1 ratio to receive "Personalized" rTMS treatment or traditional rTMS treatment in addition to routine antidepressant treatments.

Based on inclusion and exclusion criteria, after stroke depression (post-stroke depression, PSD) cases were collected and randomized into two groups: "individualized" rTMS+ drug treatment group and traditional rTMS plus traditional drug treatment group. The main indicators were the effective rate of treatment.Based on inclusion and exclusion criteria, after stroke depression (post-stroke depression, PSD) cases were collected and randomized into two groups: "individualized" rTMS+ drug treatment group and traditional rTMS plus traditional drug treatment group. The main indicators were the effective rate of treatment. The primary outcome is the measurement of 24-item Hamilton Depression Rating Scale (HAMD-24) scores, the secondary outcomes include National Institutes of Health Stroke Scale (NIHSS), Activities of Daily Living Scale (ADLs),self-rating anxiety scale(SAS). The record of the adverse reactions and sequelae during treatment and follow-up, with a view to providing a better clinical method for the treatment of PSD.

ELIGIBILITY:
Inclusion Criteria

（1） First-time ischemic stroke with clinical and MRI or CT findings of basal ganglia stroke (ICD-10-CM code 293.83[F06.32]) (3) Right-handedness (4)Clear consciousness (5)Aged 25-75 years with a recent (less than 24 months) ischemic stroke;

Exclusion Criteria

1. Aphasia or severe cognitive impairment, severe hearing impairment;
2. Contraindications of MRI scan and rTMS treatment such as pacemaker implantation; (3)Depression caused by psychoactive substances and non addictive substances;（4）Prior history of depressive disorders or major trauma within 1 year, severe depression or any other severe mental disorders;

（5）Pregnant or breast-feeding women; （6）Refusal to sign informed consent of this study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
response rate | Before treatment.1week, 2weeks, 4weeks, 8weeks after treatment
  Compare the HAMD-24 scores from baseline to the end of the treatment.the response to treatment is defined as at least a 30% reduction of the HAMD-24 total score with a final HAMD-24 score. The score decreased by more than 50% for the treatment of good results.The response rate is defined as the percentage of number of response.

SECONDARY OUTCOMES:
Neuropsychological tests results of SAS | Before treatment.1week, 2weeks, 4weeks, 8weeks after treatment
  Get the change of the result of self-rating anxiety scale (SAS) by Comparing the change of SAS scores from baseline to the end of the treatment in each group.
Neuropsychological tests results of ADLs | Before treatment.1week, 2weeks, 4weeks, 8weeks after treatment
  Get the change of the result of Activities of Daily Living Scale (ADLs) by Comparing the change of ADLs scores from baseline to the end of the treatment in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wu, M.D., Study Chair — Zhujiang Hospital
Locations (1):
- Zhujiang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broomfield NM, Quinn TJ, Abdul-Rahim AH, Walters MR, Evans JJ. Depression and anxiety symptoms post-stroke/TIA: prevalence and associations in cross-sectional data from a regional stroke registry. BMC Neurol. 2014 Oct 1;14:198. doi: 10.1186/s12883-014-0198-8. PMID 25269762
- [Background] Concerto C, Lanza G, Cantone M, Ferri R, Pennisi G, Bella R, Aguglia E. Repetitive transcranial magnetic stimulation in patients with drug-resistant major depression: A six-month clinical follow-up study. Int J Psychiatry Clin Pract. 2015;19(4):252-8. doi: 10.3109/13651501.2015.1084329. Epub 2015 Sep 23. PMID 26398527
- [Background] Damasio A, Carvalho GB. The nature of feelings: evolutionary and neurobiological origins. Nat Rev Neurosci. 2013 Feb;14(2):143-52. doi: 10.1038/nrn3403. PMID 23329161
- [Background] De Ryck A, Brouns R, Geurden M, Elseviers M, De Deyn PP, Engelborghs S. Risk factors for poststroke depression: identification of inconsistencies based on a systematic review. J Geriatr Psychiatry Neurol. 2014 Sep;27(3):147-58. doi: 10.1177/0891988714527514. Epub 2014 Apr 7. PMID 24713406
- [Background] De Ryck A, Fransen E, Brouns R, Geurden M, Peij D, Marien P, De Deyn PP, Engelborghs S. Poststroke depression and its multifactorial nature: results from a prospective longitudinal study. J Neurol Sci. 2014 Dec 15;347(1-2):159-66. doi: 10.1016/j.jns.2014.09.038. Epub 2014 Oct 2. PMID 25451004
- [Background] Dwyer Hollender K. Screening, diagnosis, and treatment of post-stroke depression. J Neurosci Nurs. 2014 Jun;46(3):135-41. doi: 10.1097/JNN.0000000000000047. PMID 24670433
- [Background] Eriksen S, Gay CL, Lerdal A. Acute phase factors associated with the course of depression during the first 18 months after first-ever stroke. Disabil Rehabil. 2016;38(1):30-5. doi: 10.3109/09638288.2015.1009181. Epub 2015 Feb 6. PMID 25655394
- [Background] Jastorff J, Huang YA, Giese MA, Vandenbulcke M. Common neural correlates of emotion perception in humans. Hum Brain Mapp. 2015 Oct;36(10):4184-201. doi: 10.1002/hbm.22910. Epub 2015 Jul 28. PMID 26219630
- [Background] Li W, Ling S, Yang Y, Hu Z, Davies H, Fang M. Systematic hypothesis for post-stroke depression caused inflammation and neurotransmission and resultant on possible treatments. Neuro Endocrinol Lett. 2014;35(2):104-9. PMID 24878979
- [Background] Narushima K, Kosier JT, Robinson RG. A reappraisal of poststroke depression, intra- and inter-hemispheric lesion location using meta-analysis. J Neuropsychiatry Clin Neurosci. 2003 Fall;15(4):422-30. doi: 10.1176/jnp.15.4.422. PMID 14627768
- [Background] Riccelli R, Passamonti L, Cerasa A, Nigro S, Cavalli SM, Chiriaco C, Valentino P, Nistico R, Quattrone A. Individual differences in depression are associated with abnormal function of the limbic system in multiple sclerosis patients. Mult Scler. 2016 Jul;22(8):1094-105. doi: 10.1177/1352458515606987. Epub 2015 Oct 9. PMID 26453680
- [Background] Robinson RG, Lipsey JR, Rao K, Price TR. Two-year longitudinal study of post-stroke mood disorders: comparison of acute-onset with delayed-onset depression. Am J Psychiatry. 1986 Oct;143(10):1238-44. doi: 10.1176/ajp.143.10.1238. PMID 3766786
- [Background] Sun N, Li QJ, Lv DM, Man J, Liu XS, Sun ML. A survey on 465 patients with post-stroke depression in China. Arch Psychiatr Nurs. 2014 Dec;28(6):368-71. doi: 10.1016/j.apnu.2014.08.007. Epub 2014 Sep 3. PMID 25457685
- [Background] Valiengo L, Casati R, Bolognini N, Lotufo PA, Bensenor IM, Goulart AC, Brunoni AR. Transcranial direct current stimulation for the treatment of post-stroke depression in aphasic patients: a case series. Neurocase. 2016;22(2):225-8. doi: 10.1080/13554794.2015.1130231. Epub 2016 Jan 8. PMID 26743441
- [Background] Wichowicz HM, Gasecki D, Landowski J, Lass P, Swierkocka M, Wisniewski G, Nyka WN, Wilkowska A. Clinical utility of chosen factors in predicting post-stroke depression: a one year follow-up. Psychiatr Pol. 2015;49(4):683-96. doi: 10.12740/PP/38439. English, Polish. PMID 26488345
- [Background] Yang S, Hua P, Shang X, Cui Z, Zhong S, Gong G, Humphreys GW. A significant risk factor for poststroke depression: the depression-related subnetwork. J Psychiatry Neurosci. 2015 Jul;40(4):259-68. doi: 10.1503/jpn.140086. PMID 25871495
- [Background] Zhao Q, Tang Y, Chen S, Lyu Y, Curtin A, Wang J, Sun J, Tong S. Early perceptual anomaly of negative facial expression in depression: An event-related potential study. Neurophysiol Clin. 2015 Dec;45(6):435-43. doi: 10.1016/j.neucli.2015.09.011. Epub 2015 Nov 18. PMID 26602972
- [Derived] Zhang X, Shi Y, Fan T, Wang K, Zhan H, Wu W. Analysis of Correlation Between White Matter Changes and Functional Responses in Post-stroke Depression. Front Aging Neurosci. 2021 Oct 11;13:728622. doi: 10.3389/fnagi.2021.728622. eCollection 2021. PMID 34707489